CLINICAL TRIAL: NCT06640894
Title: Power2Walk: The Impact of Functional Power Training on Participation and Activity in Children With Cerebral Palsy - A Randomized Controlled Trial
Brief Title: Power2Walk: The Impact of Functional Power Training on Participation and Activity in Children With Cerebral Palsy.
Acronym: Power2Walk
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Amsterdam UMC, location VUmc (Other)
Collaborators: Netherlands Brain Foundation (Other); Koninklijk Nederlands Genootschap voor Fysiotherapie (Unknown); De Phelps Stichting voor Spastici (Unknown); Reade Rheumatology Research Institute (Other); Adelante, Centre of Expertise in Rehabilitation and Audiology (Other); Heliomare (Unknown); Merem (Unknown); Revant (Unknown); Revalidatie Friesland (Unknown); Roessingh (Unknown); Treant Zorggroep (Unknown); Johanna Kinderfonds (Unknown)
Responsible Party: Principal Investigator, Rijk Dersjant, Coordinating investigator, VU University of Amsterdam
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NL85905.018.23; 2024.0022 (Other: METC Amsterdam UMC)
Record Dates: First submitted 2024-08-19; First posted 2024-10-15 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Cerebral Palsy, Spastic
Keywords: Cerebral palsy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Intervention Model Description: A single-blind randomized controlled parallel trial with a 24 week follow-up.
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (MegaPower training) (Experimental): MegaPower training is a twelve-week long functional power training program in which children will perform functional power training three times a week together with a personal trainer. During the intervention, training volume will be influenced by training weight, velocity of movement, and amount of repetitions. The training program has the following characteristics:
  1. (Weighted) functional exercises like walking, running, and walking stairs.
  2. High velocity movements.
  3. Progressive overload.
  Prior to and during the training, a physiotherapist makes a personalized participation plan for the child. This plan is used to tackle participation barriers related to their goal (not directly related to mobility; e.g. beliefs or behaviours) encountered by the child (e.g. involving parents, a sports consultant, a psychologist).
  Both at twelve and twenty-four weeks during the follow-up, parent and child will visit again to measure whether the effects on participation are long-lasting.
  Interventions: Other: MegaPower training
- Control (Usual Care) (Active Comparator): The control group will receive their usual care for twelve weeks (non-intervention group). This usual care consists of physiotherapy appointments, for example.
  Interventions: Other: Usual Care

INTERVENTIONS:
Other: MegaPower training — See arm/group descriptions
  Arms: Intervention (MegaPower training)
Other: Usual Care — See arm/group descriptions
  Arms: Control (Usual Care)

SUMMARY:
Rationale: Children with cerebral palsy (CP) experience limitations in walking ability due to functional motor impairments caused by neurodevelopmental damage during fetal or early child development. Due to these motor impairments, children with CP struggle to keep up with typically developing peers when participating in physical and/or social activities. Consequently, the development of these children may be hampered. Recently, functional power training (FPT) emerged as a potentially successful supplementary treatment method to improve participation in children with CP. It is understood that FPT is more effective than progressive resistance training in improving walking ability and endurance, and thereby better supports participation in ambulatory children with CP. Nevertheless, high-level scientific evidence underpinning the efficacy of FPT on these parameters in ambulant children with CP is still lacking. The investigators hypothesize that FPT effectively helps accomplish patient-tailored participation and activity goals in ambulant children with CP.

Objective: This study aims to investigate whether twelve weeks of FPT (MegaPower training) effectively accomplish patient-tailored participation and activity goals in ambulant children with CP, when compared to their usual care. Additionally, the goal is to investigate i) whether MegaPower training improves walking ability, aerobic endurance, and anaerobic capacity; ii) what factors best identify which ambulant children with CP benefit most from twelve weeks of MegaPower training; iii) to what extend the MegaPower training was implemented as intended in the participating study centers?, and iv) whether the effects of the MegaPower training are maintained after 12 and 24 weeks of follow-up.

Study design: A single-blind randomized controlled parallel trial with a 24 week follow-up. During the follow-up, the control group will also receive MegaPower training.

Study population: Ambulant children with cerebral palsy or a related non-progressive disorder between the ages of 4 - 12.

Intervention: One group will receive twelve weeks of FPT (MegaPower training), whilst the other group will receive twelve weeks of usual care (control group).

Main study parameters/endpoints: Accomplishment of patient-tailored participation and activity goals, measured through Goal Attainment Scaling.

DETAILED DESCRIPTION:
Children with cerebral palsy (CP) experience limitations in walking ability due to functional motor impairments caused by neurodevelopmental damage during fetal or early child development that may result in spasticity, dyskinesia, or ataxia. Due to these motor impairments, children with CP struggle to keep up with typically developing peers when participating in physical and/or social activities. Yet, participation is a key factor in child development, mainly because it is instrumental in enhancing mental well-being through building friendships, developing a personal identity, optimizing physical growth, and increasing motor control. Earlier studies concluded that children with CP are indeed at an elevated risk for reduced physical activity and participation. Consequently, the development of these children may be hampered. Therefore, targeted interventions that increase physical activity and participation are essential for supporting the general development of children with CP. A large number of treatments have been developed for children with CP, ranging from pharmacological agents that manage tone to invasive surgical interventions. Whilst many of these treatments effectively improve motor control, very few address the underlying fatigue that is typically seen in these children, which causes a vicious cycle of reduced physical fitness, early onset of fatigue, and decreased physical activity levels. This decline in physical fitness is ultimately detrimental to participation, and therefore a wide variety of exercise-related treatment options are being explored to improve motor control, physical fitness, and participation.

Recently, functional power training (FPT) emerged as a potentially successful supplementary treatment method to improve participation in children with CP. This type of strength training combines high velocity movements with progressive resistance to mimic and train the demands of playing activities like playground running and sprinting in games and sports. Indeed, a previous double-baseline study indicated that FPT improves physical fitness, muscle strength, activity, and participation in ambulatory children with CP. This is unlike progressive resistance training (PRT), which increases muscle strength but not walking ability, anaerobic capacity, and ultimately participation. This discrepancy is likely explained by the functional nature of FPT, which specifically trains activities of daily living and not only muscle strength. Moreover, power training may be more effective than strength training as power training incorporates high intensity, explosive-like contractions that are required in daily living situations. Consequently, FPT is more effective than PRT in improving walking ability, thereby better supporting participation in ambulatory children with CP. Nevertheless, high-level scientific evidence underpinning the efficacy of FPT on walking ability, aerobic endurance, anaerobic capacity, and participation in ambulant children with CP is still lacking. Furthermore, it remains unclear what predictive factors best identify which children with CP benefit most from FPT. Additionally, it remains unknown whether the potential benefits of FPT on walking ability, aerobic endurance, anaerobic capacity, and participation in children with CP are maintained when FPT is discontinued.

ELIGIBILITY:
Inclusion Criteria:

* Children with cerebral palsy or a related non-progressive disorder between the ages of 4 to 12.
* Gross Motor Function Classification System (GMFCS) level I - III.
* Parents and/or children have a treatment question related to participation of the child.

Exclusion Criteria:

* Participants that suffer from a progressive neurological disorder.
* Treatment with botulinum toxin and/or serial casting in lower extremities planned during the study period.
* Treatment with botulinum toxin in the twelve weeks prior to participation in the study.
* Treatment with serial casting in the three weeks prior to participation in the study.
* Children that underwent a selective dorsal rhizotomy twelve months prior to participation in the study.
* Children that underwent orthopedic surgery on their lower extremities in the 12 months before participation in the study.
* Children that have received MegaPower training in the last 4 months before participation in the study.
* Children for whom walking is not their preferred method of locomotion (yet).

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 66 (Estimated)
Dates: Start 2024-07-19 (Actual); Primary Completion 2027-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Goal Attainment (Goal Attainment Scaling) | Baseline (t = 0 weeks); t = 12 weeks, t = 24 weeks, t = 36 weeks.
  Goal Attainment Scaling (GAS) is a method used to measure the achievement of individual goals in a structured and quantitative manner. It is commonly used in clinical and educational settings to evaluate progress and outcomes. Each goal is scaled on a six-point scale, ranging from -3 to +2:
  Goal Attainment Scaling endpoints will be formulated according to SMART-principles to standardize results.

SECONDARY OUTCOMES:
Mobility Questionnaire 28 (MobQues28) | Baseline (t = 0 weeks); t = 12 weeks, t = 24 weeks, t = 36 weeks.
  The MobQues28 is a parent-reported mobility questionnaire used in cerebral palsy research that assesses gait-related function across different domains of the International Classification of Functioning, Disability and Health (ICF) developed for ambulant children with CP.
Gait Outcomes Assessment List (GOAL) | Baseline (t = 0 weeks); t = 12 weeks, t = 24 weeks, t = 36 weeks.
  The GOAL is a parent-reported mobility questionnaire that assesses gait-related function across different domains of the ICF and is developed for ambulant children with CP. The GOAL is a more comprehensive and better standardized version of the MobQues28. However, since our study population is based off expected differences in the MobQues28 (since data for the GOAL on this subject does not exist yet), both questionnaires are included.
Harter's Self-Perception Profile for Children | Baseline (t = 0 weeks); t = 12 weeks, t = 24 weeks, t = 36 weeks.
  Harter's Self-Perception Profile for Children (HSPPC) is a psychological assessment tool designed to measure self-concept in children. Children will be assessed on the domains of social competence, athletic competence, and global self-worth.
Physical activity (accelerometer) | Baseline (t = 0 weeks); t = 12 weeks
  Physical activity will be measured over a 7-day period using a wearable accelerometer that participants will have to carry for seven days. The accelerometer picks up accelerations of the body and can accurately estimate physical (in)activity accordingly. The accelerometer does not have an interface and does not save any personal data.
Sleep (accelerometer) | Baseline (t = 0 weeks); t = 12 weeks
  Sleep will be measured over a 7-day period using a wearable accelerometer that participants will have to carry for seven days. The accelerometer picks up accelerations of the body and can estimate sleep duration and quality. The accelerometer does not have an interface and does not save any personal data.
Body composition (bioelectrical impedance analysis) | Baseline (t = 0 weeks); t = 12 weeks, t = 24 weeks, t = 36 weeks.
  Body composition; measured using bioelectrical impedance analysis (BIA). BIA is a method to assess body composition based on the resistance of different tissue types against an unnoticeable electric pulse through the body, since fat mass and fat free mass have a different conductivity.
Walking speed (1-minute walk test) | Baseline (t = 0 weeks); t = 12 weeks, t = 24 weeks, t = 36 weeks.
  The 1-minute walk test is a physical test that measures walking speed. The child is asked to walk as quickly as possible around a measured track for a period of one minute. The distance walked within 1 minute is measured and recorded.
Aerobic endurance (shuttle run test) | Baseline (t = 0 weeks); t = 12 weeks, t = 24 weeks, t = 36 weeks.
  The shuttle run test is a physical test that measures aerobic endurance. Children walk or run at a set incremental speed between two markers that are placed ten meters apart. These walks/runs are coordinated by a recorded CD that plays a sound at pre-determined intervals. Children have to keep up with the speed of these intervals and are measured by the level they reached. Different validated tests will be used for children of different GMFCS levels.
Anaerobic capacity (muscle power sprint test). | Baseline (t = 0 weeks); t = 12 weeks, t = 24 weeks, t = 36 weeks.
  The Muscle Power Sprint Test is a physical test that measures anaerobic capacity. Children have to perform a fifteen meter sprint as fast as possible, repeated six times with ten seconds of rest in between. Their score will be presented in mean and peak power (force * speed).
Dietary intake (3-day food record) | Baseline (t = 0 weeks).
  Dietary intake at baseline; measured using a 3-day food record in which parents have to track the nutritional intake of their child during two week days and one weekend day.
Process evaluation | Through study completion. An average of 2 years.
  A process evaluation will be employed to monitor and document program implementation. With this information, the goal is to evaluate to what extend the MegaPower training was implemented as intended in the participating study centers. This allows us to understand the relationship between specific program elements and program outcomes. The framework by Saunders et al., describing five components of process evaluation will be used. The methods proposed contains questionnaires, report and registration forms, interviews, and focus groups. As a part of this process evaluation, parents will also be asked to fill out a questionnaire about whether their child is happy with the care they received.
Age | Baseline (t = 0 weeks)
  Age (years and months) at start of study.
Height (cm) | Baseline (t = 0 weeks); t = 12 weeks, t = 24 weeks, t = 36 weeks.
Weight (kg) | Baseline (t = 0 weeks); t = 12 weeks, t = 24 weeks, t = 36 weeks.
Gender (male/female/other) | Baseline (t = 0 weeks)
GMFCS level (I, II, or III) | Baseline (t = 0 weeks)
  The mobility and gross motor skills of people with cerebral palsy are categorized into five different levels using a tool called the Gross Motor Function Classification System (GMFCS).
Type of cerebral palsy | Baseline (t = 0 weeks)
  Spastic/dyskinetic/ataxic/unilateral/bilateral/hemiplegia/diplegia/quadriplegia/other.
Type of education (regular/special) | Baseline (t = 0 weeks)
Education level of parent(s) | Baseline (t = 0 weeks)
Use of ankle-foot orthoses (yes/no) | Baseline (t = 0 weeks)
Participation in sports | Baseline (t = 0 weeks)
  Do the child and the family of the child participate in any sports? And if so, how many times a week?

CONTACTS AND LOCATIONS:
Overall Officials: Annemieke I. Buizer, prof. dr., Principal Investigator — Amsterdam UMC
Locations (10):
- Netherlands (10):
  - Treant Zorggroep, Emmen, Drenthe
  - Merem, Almere Stad, Flevoland
  - Adelante zorggroep, Valkenburg, Limburg
  - Revant, Breda, North Brabant
  - Reade, Amsterdam, North Holland
  - Heliomare, Heemskerk, North Holland
  - Merem, Hilversum, North Holland
  - Roessingh, Enschede, Overijssel
  - Revalidatie Friesland, Beetsterzwaag, Provincie Friesland
  - Revant, Goes, Zeeland

IPD SHARING:
Plan to Share IPD: No